CLINICAL TRIAL: NCT06602570
Title: The Mosaic Brain: a New Diagnostic Approach in Focal Epilepsies
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23BM09
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy Intractable; Epilepsy in Children
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Overall, this observational cohort study aims to:

1. Improve our understanding of the genetic architecture of childhood focal epilepsies.
2. Develop a liquid biopsy of cerebrospinal fluid (CSF) and assess feasibility to detect cerebral mosaicism using cell-free DNA (cfDNA) analysis and evaluate its performance against brain tissue on the panel testing.
3. Develop a methodology to use trace tissue from Stereoelectroencephalography (SEEG) DNA and assess feasibility to detect cerebral mosaicism and evaluate its performance against brain tissue on the panel testing.

3. Validate the use of the liquid biopsy and SEEG trace tissue for use in the English National Health Service clinical services and share with other Genomic Laboratory Hubs.

DETAILED DESCRIPTION:
Epilepsy is characterised by recurrent epileptic seizures, and is the most common brain disease affecting children, significantly reducing their quality of life. Understanding the cause of epilepsy is key, as it can help doctors to identify the most effective treatment. This is an urgent issue as 30% of all children with epilepsy do not respond to currently available treatments.

In some children, seizures can start in an area of abnormal brain structure which can be removed with epilepsy surgery.

We see 150 children a year with epilepsy suspected to be caused by a brain lesion. As part of their evaluation, we do genetic testing in blood, as we know that changes in their DNA (mutations) can cause epilepsy in 30-40% of children.

It is now known that mutations are found in some areas of brain responsible for seizures but these are not present in the blood. This is mosaicism, when genetic variation affects only a subgroup of cells or tissues in an individual. Understanding these genetic changes in the brain tissue will help us understand how epilepsy starts and may help us design new treatments. Recently, we designed a new genetic test to pick up these mosaic mutations in brain tissue. However, current methods to detect mosaicism require the use of brain tissue, which limits testing to those children who qualify for surgery.

To expand testing to more children, without the need for surgery, we want to focus our work in using alternative samples, such as cell-free DNA cerebrospinal fluid (CSF) and trace-tissue DNA from trace cells collected from Stereoelectroencephalography (SEEG) electrodes.

We aim to further our understanding of brain mosaicism in epilepsy, using the current available tests, as well as aim to increase access to testing by developing methods to use samples collected using less invasive and pre-surgical methods.

ELIGIBILITY:
Inclusion Criteria:

* Children in the epilepsy surgery pathway at Great Ormond Street Hospital (GOSH) with a clear or suspected MRI lesion.
* All children undergoing SEEG at GOSH. Children for which consent was obtained from themselves or, if appropriate, from their legal representatives.
* Children in whom there are no clinical contraindication to having a lumbar puncture procedure pre-surgery.
* Both sexes.
* Under the age of 18.

Exclusion Criteria:

* Children that although undergoing epilepsy treatment or testing for an ischaemic lesion.
* Children with malignant brain tumours.
* Children in whom there are contraindications to performing a lumbar puncture procedure.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: - Children in the epilepsy surgery service at GOSH.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Measure concordance of genetic results for brain mosaicism testing between brain tissue and alternative samples. | 24 months

SECONDARY OUTCOMES:
Present and compare DNA quality metrics from the several samples types using different methodologies and select the methods yielding better sample quality. | 24 months
Measure concordance between variant allele frequency (VAF) from brain tissue mosaic genetic testing and VAF calculated using alternative samples. | 24 months
Present and compare mosaic genetic variability results between alternative samples (cell-free DNA and trace tissue DNA) and peripheral blood DNA. | 24 months
Present descriptive statistics detailing changes to patient management and genetic counselling directly resulting from a genetic mosaic diagnosis. | 24 months